CLINICAL TRIAL: NCT07317102
Title: Omnipod-5 A French Prospective Multicentric Study in Real World (Optimal-B)
Status: Not yet recruiting | Type: Observational
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Optimal-B
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetes; Type 1 Diabetes; Diabetes Mellitus
Keywords: Omnipod; Automated Insulin Delivery; Post-market Registry
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Omnipod 5 User: Participation of each patient begins at inclusion and continues until the end-of-study visit, 12 months (± 1 month) following first initiation of automated mode of the Omnipod 5 System
  Interventions: Device: Omnipod 5

INTERVENTIONS:
Device: Omnipod 5 — The Omnipod 5 Automated Insulin Delivery System (Omnipod 5 System) is a tubeless insulin pump with a mono-hormonal insulin delivery system designed to deliver U-100 insulin subcutaneously for the management of type 1 diabetes in people aged 2 years and older who require insulin.
  The Omnipod 5 System is intended to function as an automated insulin delivery system when used with compatible Continuous Glucose Monitoring (CGM) systems.

SUMMARY:
The purpose of this postmarket clinical investigation is to evaluate the levels of glycemic control, quality of life, and satisfaction, as well as the patient experience, and acute diabetes complication rates provided by the Omnipod 5 Automated Insulin Delivery System (referred to as the Omnipod 5 System) in a real-world setting.

DETAILED DESCRIPTION:
Twelve-month, real-world, non-interventional, prospective follow-up of adult and pediatric patients aged more than 2 years old, prescribed the commercially available FreeStyle Libre 2 Plus configuration of the Omnipod 5 Automated Insulin Delivery System in France.

OPTIMAL-B study (Omnipod 5 - A French Prospective Multicentric Study in Real World), aims to provide the requisite real-world data on the glycemic control, quality of life, safety, and device usage profiles of users of the Omnipod 5 System during the 12 months after starting using Omnipod 5 in automated mode.

ELIGIBILITY:
Inclusion Criteria:

* Patient with T1D aged ≥ 2 years.
* Patient prescribed, less than a year ago, a commercially available confi guration of the Omnipod 5 System using a FreeStyle Libre 2 Plus sensor.
* Patient has never used the Omnipod 5 System prior to inclusion.
* Patient has not objected to the use of their personal data for this study.
* Patient or legal guardian has an email address and mobile phone number.
* Patient (and legal guardians if the patient is a minor) is able to understand study information and Non-Opposition form.
* Patient (and legal guardians if the patient is a minor) is able to understand and complete questionnaires in French.
* Patient is covered by the local social security system

Exclusion Criteria:

* Patient is currently pregnant.
* Patient presents an allergy to the materials of the Omnipod 5 System (patch, cannula, CGM).
* Patient is unable to be followed by the same investigation site for the duration of the study or is unwilling or unable to maintain contact with the healthcare professional.
* Patient is already participating in a clinical trial or in another study precluding their participation in other studies.
* Adult under guardianship, curatorship or tutorship.
* Adult otherwise deprived of liberty.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population contains patients (age ≥ 2 years) with T1DM initiating a commercially available configuration of the Omnipod 5 System using a FreeStyle Libre 2Plus in France.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of time in the 70 - 180 mg/dL range | Change in percentage of time in specified range between Baseline and 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control

SECONDARY OUTCOMES:
Percentage of time in the 70 - 180 mg/dL range | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Percentage of time in the 70 - 140 mg/dL range | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Percentage of time below 54 mg/dL | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Percentage of time below 70 mg/dL | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Percentage of time above 180 mg/dL | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Percentage of time above 250 mg/dL | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Glucose Management Indicator (GMI) | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Glycemic Risk Index (GRI) | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Coefficient of variation (CV) | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
Mean glucose | Up to 12-months following first initiation of automated mode
  Glucose metric from continuous glucose monitoring system to assess glucose control
HbA1c Level (if available) | Up to 12-months following first initiation of automated mode
  Blood test to assess glucose control
Percentage of patients with ≥ 70% | Up to 12-months following first initiation of automated mode
  Assess the achievement of CGM-based consensus targets
Percentage of patients with < 4% | Up to 12-months following first initiation of automated mode
  Assess the achievement of CGM-based consensus targets
Percentage of patients with < 1% | Up to 12-months following first initiation of automated mode
  Assess the achievement of CGM-based consensus targets
Percentage of patients with GMI ≤ 7% | Up to 12-months following first initiation of automated mode
  Assess the achievement of CGM-based consensus targets
Percentage of patients with CV ≤ 36% | Up to 12-months following first initiation of automated mode
  Assess the achievement of CGM-based consensus targets
Percentage of patients achieving combinations of previous CGM-based consensus targets | Up to 12-months following first initiation of automated mode
  Assess the achievement of CGM-based consensus targets
EuroQoL 5-dimension 5-level questionnaire | At inclusion and 6 and 12 months following first initiation of automated mode
  Assess patients' general quality of life
Patients aged ≥ 18 years: Diabetes Quality of Life - Brief Clinical Inventory | At inclusion and 6 and 12 months following first initiation of automated mode
  Assess patients' diabetes-specific quality of life
Patients aged 10-17 years: Diabetes Quality of Life for Youth scale - Short Form (DQOLY-SF) | At inclusion and 6 and 12 months following first initiation of automated mode
  Assess patients' diabetes-specific quality of life
Insulin Delivery System Rating Questionnaire (IDSRQ) interference sub-score | At inclusion and 6 and 12 months following first initiation of automated mode
  Assess the interference of the Omnipod 5 System with patients' daily lives
Patients aged ≥ 18 years: Diabetes Treatment Satisfaction Questionnaire, status version(DTSQs) | At inclusion and 6 and 12 months following first initiation of automated mode
  Assess patients' satisfaction with the Omnipod 5 System
Patients aged 13-17 years: Diabetes Treatment Satisfaction Questionnaire, status version -Teens (DTSQs - Teen) | At inclusion and 6 and 12 months following first initiation of automated mode
  Assess patients' satisfaction with the Omnipod 5 System
Patients aged 2-12 years: Diabetes Treatment Satisfaction Questionnaire, status version -Parent (DTSQs - Parent) | At inclusion and 6 and 12 months following first initiation of automated mode
  Assess patients' satisfaction with the Omnipod 5 System
Pediatric quality of life questionnaire (animated emoji scale - ad hoc) | At inclusion and 6 and 12 months following first initiation of automated mode
  Assess pediatric patients' quality of life with the Omnipod 5 System
Percentage of time using the System in automated mode | 12 months following first initiation of automated mode
  Describe System use
Percentage of time using the System in manual mode | 12 months following first initiation of automated mode
  Describe System use
Percentage of time using "Activity" feature | 12 months following first initiation of automated mode
  Describe System use
Total daily dose of insulin | 12 months following first initiation of automated mode
  Describe System use
Number of boluses per day | 12 months following first initiation of automated mode
  Describe System use
Targets used by patients | 12 months following first initiation of automated mode
  Describe System use
Bolus/Basal distribution | 12 months following first initiation of automated mode
  Describe System use
Incidence of severe hypoglycemia | 6 months prior to switching to Omnipod 5 and over the 12 months following first initiation of automated mode
  Assess the incidence and type of acute metabolic complications
Incidence of diabetic ketoacidosis | 6 months prior to switching to Omnipod 5 and over the 12 months following first initiation of automated mode
  Assess the incidence and type of acute metabolic complications
Unscheduled hospitalizations for diabetes or diabetes complications | 6 months prior to switching to Omnipod 5 and over the 12 months following first initiation of automated mode
  Assess the incidence and type of acute metabolic complications
Percentage of patients still using the Omnipod 5 System at the end of study follow-up | 12 months following first initiation of automated mode
  Assess the rate at which patients stop using the Omnipod 5 system
Reasons for having stopped using the Omnipod 5 System | 12 months following first initiation of automated mode
  Assess the rate at which patients stop using the Omnipod 5 system

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Riveline, MD, PhD, Principal Investigator — Centre Universitaire du Diabète et ses complications Hôpital Lariboisière
Locations (22):
- France (22):
  - CHU Angers, Angers
  - CHU Besançon - Hôpital de Jean Minjoz, Besançon
  - APHP Hopital Avicenne, Bobigny
  - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHU Bordeaux - Hôpital St-André, Bordeaux
  - CHU Brest - Hôpital de la Cavale Blanche, Brest
  - Hôpital Femme Mère Enfant, Bron
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CIRDIA, Dijon
  - CHU Dijon - Hôpital François Mitterrand, Dijon
  - GH La Rochelle-Ré-Aunis - Hôpital Saint Louis, La Rochelle
  - APHP Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Institut de Diabétologie et de Nutrition du Centre, Mainvilliers
  - Fondation Ambroise Paré - Hôpital Européen de Marseille, Marseille
  - CHU Montpellier - Hôpital Lapeyronie, Montpellier
  - Institut Saint Pierre, Palavas-les-Flots
  - APHP Hôpital Lariboisière, Paris
  - APHP Hopital Robert Debré, Paris
  - CH Périgueux, Périgueux
  - Clinique Saint Jean de Védas, Saint-Jean-de-Védas
  - CHRU Strasbourg, Strasbourg
  - CHU Tours, Tours